CLINICAL TRIAL: NCT00655031
Title: A Placebo Controlled, Randomized, Double Blind Pilot Study to Evaluate the Use of Pomegranate Concentrate (POMx) for the Prevention of Experimental Rhinovirus Infection in Human Subjects
Brief Title: Trial to Evaluate the Use of Pomegranate Concentrate (POMx) for the Prevention of Experimental Rhinovirus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: POM Wonderful LLC (Industry)
Responsible Party: Mark Dreher / Vice President, Scientific and Regulatory Affairs, POM Wonderful LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A004
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Common Cold
Keywords: Punicaceae; Pomegranate
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Pomegranate concentrate (POMx)
  Interventions: Dietary Supplement: Pomegranate Concentrate (POMx)
- 2 (Placebo Comparator): Fruit flavored juice low in antioxidants
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pomegranate Concentrate (POMx) — 3.3 oz bottle containing antioxidants equivalent to 8 oz of pomegranate juice taken once daily for 7 days prior to infection and for 4 days after.
  Arms: 1
Dietary Supplement: Placebo — 3.3 oz bottle containing fruit flavored juice low in antioxidants taken once daily for 7 days prior to infection and for 4 days after.
  Arms: 2

SUMMARY:
Pomegranate has a long history of use in folk medicine. There is vast data on the health benefits of pomegranate fruit and juice. Multiple studies have established the strong antioxidative effects of pomegranate polyphenols (primarily the ellagitannin punicalagin) and their health effects. A vast number of animal and human clinical studies have provided evidence on effect of pomegranate products on reducing symptoms of common cold, reducing blood pressure, improving endothelial function, anti-tumor activity, and its anti-atherosclerotic activity. This study will evaluate the protective effect of a pomegranate concentrate (POMx) in decreasing the incidence and duration of the common cold among healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoker
* No recent history of respiratory disease

Exclusion Criteria:

* Serum positive for rhinovirus
* Pregnant or breastfeeding
* Recent immunization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who become infected in the active treatment group compared with the proportion of subjects who become infected in the placebo treatment group. | Days 1-5

SECONDARY OUTCOMES:
Comparison of symptom scores in the treatment groups | Days 1-5
Determination of effects of treatment on immune function. | Days 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Turner, MD, Principal Investigator — University of Virginia
Locations (3):
- United States (3):
  - Accelovance Inc., Huntsville, Alabama
  - Accelovance Inc, Melbourne, Florida
  - University of Virginia School of Medicine, Charlottesville, Virginia